CLINICAL TRIAL: NCT05576298
Title: Pharmacokinetics, Pharmacodynamic, Safety and Immunogenicity Characteristics of Insulin Degludec Injection (RD15003) and Insulin Degludec Injection ( Tresiba®）in Healthy Subjects: a Phase I Single-center, Randomized, Open-label, Single-dose, Cross-over Clinical Study
Brief Title: A Clinical Study Comparing the Pharmacokinetics and Pharmacodynamic Characteristics of Insulin Degludec Injection (RD15003) and Insulin Degludec Injection (Tresiba®) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RD15003-P-01
Record Dates: First submitted 2022-09-14; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR sequence (Experimental): Experimental:Insulin degludec injection (RD15003)+Tresiba Subjects receive Insulin degludec injection(RD15003) in the first cycle and Tresiba in the second cycle.
  Interventions: Biological: Insulin degludec injection, RD15003; Biological: Insulin degludec, Tresiba
- RT sequence (Experimental): Experimental:Tresiba+Insulin degludec injection (RD15003) Subjects receive Insulin Tresiba in the first cycle and degludec injection(RD15003) in the second cycle.
  Interventions: Biological: Insulin degludec injection, RD15003; Biological: Insulin degludec, Tresiba

INTERVENTIONS:
Biological: Insulin degludec injection, RD15003 — single dose, s.c. injection
Biological: Insulin degludec, Tresiba — single dose, s.c. injection

SUMMARY:
To evaluate the single-dose subcutaneous injection of insulin degludec injection (Tresiba®) listed by Novo Nordisk in China as a reference drug, the insulin degludec injection provided by Dongguan Dongyang Sunshine Biopharmaceutical R&D Co., Ltd. (RD15003) pharmacokinetics and pharmacodynamic characteristics in healthy subjects, and then to evaluate the bioequivalence of test drugs and control drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the trial, and sign the informed consent form, and be able to complete the trial in accordance with the requirements of the plan;
2. When signing the informed consent form, healthy subjects aged 18-45 (including the cut-off value) are not limited to males and females;
3. At the time of screening, male weight > or = 50 kg, female weight > or = 45 kg, body mass index (BMI) > or = 19.0 and < or = 26.0 kg/m2;
4. After medical history inquiry, there is no clinically significant heart, liver, kidney, digestive tract, nervous system disease, and metabolic abnormality history;
5. Vital signs, physical examination, laboratory examination and/or ECG, chest X-ray examination results are normal or abnormal, but the investigator judges that they have no clinical significance;
6. Normal glucose tolerance [fasting blood glucose (FPG) <6.1 mmol/L, and oral glucose tolerance test (OGTT) 2 h postprandial blood glucose <7.8 mmol/L];
7. Insulin release test (IRT) results are normal or abnormal, but the investigator judges that it has no clinical significance;
8. Have good venous conditions, so that blood collection channels can be established according to the research plan;
9. There was no birth plan during the study period and promised to use reliable contraceptive measures throughout the study period until 4 weeks after the last administration of the trial drug.

Exclusion Criteria:

1. Have a history of hypoglycemia within 3 months before screening;
2. Those who have taken any prescription drugs, Chinese herbal medicines, over-the-counter drugs (except for subjects with occasional and restricted use of paracetamol), and health care products (except routine supplementary vitamins and calcium) within 4 weeks before administration;
3. During screening, the test results of human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or Treponema pallidum antibody were positive;
4. Have a history of malignant tumors before screening;
5. Participated in any drug or device clinical research within 3 months before screening (the definition of participation: refers to random or receiving experimental drugs or devices);
6. Blood donation > or = 400 mL within 3 months before administration, or blood loss > or = 400 mL due to any reason;
7. People who are known to be allergic to the test drug or its excipients;
8. People who drink regularly within 3 months before administration, that is, drink more than 21 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcoholic spirits or 150 mL of wine), or those who have a positive alcohol breath test ;
9. Those who have a positive urine drug screening;
10. Positive anti-insulin antibody during the screening period;
11. Female subjects who are breastfeeding, or women who have a positive blood pregnancy test during the screening period;
12. Those who smoked more than 10 cigarettes per day within 3 months before the administration, or failed to comply with the ban on smoking during the trial period;
13. There are any factors considered by the researcher to be unsuitable for participating in the research;
14. If during the period of new coronary pneumonia, the investigator decided to conduct relevant tests for the new coronavirus according to the requirements of the Sichuan Provincial Health Commission and West China Hospital of Sichuan University at the time of the trial, and the abnormal results have clinical significance.

Ages: 18 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to 24 hours | 24 hours after injection
  AUC0-24h
Area under the glucose infusion rate curve from administration to end of clamp from time zero to 24 hours | 24 hours after injection
  GIR-AUC0-24h

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to 12 hours | 12 hours after injection
  AUC0-12h
Area under the glucose infusion rate curve from administration to end of clamp from time zero to 12 hours | 12 hours after injection
  AUCGIR0-12h
Safety evaluation | Up to 24 weeks
  Incidence of adverse events
Area under the plasma concentration-time curve from time 12 hours to 24 hours | 12-24 hours after injection
  AUC12-24h
Area under the plasma concentration-time curve from time zero to t | 120 hours after injection
  AUC0-t
Area under the glucose infusion rate curve from administration to end of clamp from time 12 hours to 24 hours | 12-24 hours after injection
  AUCGIR, 12-24h
Maximum glucose infusion rate | 24 hours after injection
  GIRmax

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China